CLINICAL TRIAL: NCT01040897
Title: Addressing Health Literacy and Numeracy to Prevent Childhood Obesity
Acronym: GreenLight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Miami (Other); University of North Carolina, Chapel Hill (Other); New York University (Other); Stanford University (Other); Duke University (Other)
Responsible Party: Principal Investigator, Russell Rothman, Associate Professor, Internal Medicine & Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HD059794-01 (NIH); NCT03370445 (obsolete NCT alias)
Record Dates: First submitted 2009-12-28; First posted 2009-12-30 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Obesity Prevention
Keywords: Obesity prevention; Health Literacy; Health Communication
MeSH Terms: interventions — Health Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Control Arm (Active Comparator): At Active Comparative Sites, Pediatric Residents will be trained to address injury prevention issues using The Injury Prevention Program (TIPP) approach
  Interventions: Behavioral: Injury Prevention Arm
- Health Communication and Obesity Prevention (Experimental): Pediatric Residents will be training in effective health communication skills and given a toolkit of literacy/numeracy sensitive educational materials to use with families with children age 2 months to18 months during each well child visit
  Interventions: Behavioral: Health Communication and Obesity Prevention

INTERVENTIONS:
Behavioral: Health Communication and Obesity Prevention — Pediatric residents will be training in effective health communication skills and given a literacy/numeracy sensitive toolkit (GreenLight) to use with parents during all well child visits from 2 months to 18 months.
  Arms: Health Communication and Obesity Prevention
Behavioral: Injury Prevention Arm — Pediatric residents will be trained to address injury prevention using the American Academy of Pediatrics (AAP) TIPP materials.
  Arms: Active Control Arm

SUMMARY:
In 2003, Surgeon General Richard Carmona suggested that low health literacy is "one of the largest contributors to our nation's epidemic of overweight and obesity." Over 26% of preschool children are now overweight or obese, and children who are overweight by age 24 months are five times as likely as non-overweight children to become overweight adolescents. The aim of the study is to assess the efficacy of a low-literacy/numeracy-oriented intervention aimed at teaching pediatric resident physicians to promote healthy family lifestyles and prevent overweight among young children (age 0-2) and their families in under-resourced communities.

DETAILED DESCRIPTION:
In 2003, Surgeon General Richard Carmona stated that low health literacy was "one of the largest contributors to our nation's epidemic of overweight and obesity." This assertion is supported by recent studies which have found that low health literacy or numeracy is associated with poorer caregiver breastfeeding knowledge, incorrect mixing of infant formula, difficulty understanding food labels and portion sizes, and higher Body Mass Index (BMI) in adults and children. Of particular concern is the impact of the obesity epidemic on our youngest children. Over 26% of preschool children are now overweight (BMI≥85%) or obese (BMI≥95%) (based on 2007 Health and Human Services/Centers for Disease Control Expert Panel definitions). Rates of obesity in preschool children have doubled over the past decade, with the highest increases among low income and minority children-- the same communities most affected by low health literacy.

To date, clinical efforts to prevent or treat childhood obesity have had limited efficacy. Efforts need to start early, because children who are overweight by age two are five times as likely to become overweight adolescents, and subsequently at higher risk for obesity-related complications including early-onset Type-2 Diabetes and cardiovascular disease. No published clinical studies have rigorously addressed obesity prevention prior to age 2 with a specific low-literacy and numeracy focus. Addressing caregiver health literacy in early childhood is an innovative strategy to promote healthy nutrition and activity among these families and prevent unhealthy weight gain across the child's life, which would have great public health significance by preventing both child and adult chronic illness.

The proposed study is a multi-site randomized, controlled trial to assess the efficacy of a low-literacy/numeracy-oriented intervention designed to promote healthy family lifestyles and to prevent early childhood obesity. The intervention will be delivered through pediatric resident physicians in primary care settings in under-resourced communities. Four academic medical centers will be randomized: Vanderbilt University, the University of Miami, the University of North Carolina at Chapel Hill, and New York University. Two centers will receive the intervention, while the other two centers will receive an active control. At each site, a cohort of 250 English- or Spanish-speaking caregiver-child dyads will be enrolled and followed from the child's 2 month well-child visit through the 24-month well-child visit. The intervention will include a low-literacy-oriented toolkit for pediatric residents to use with families and clear health communication training for the pediatric residents. At control sites, pediatric residents will provide "usual care" with respect to lifestyle counseling, but they will also receive an injury-prevention education program to act as an attention control. The primary hypotheses are that the intervention will improve family dietary and physical activity behaviors and that it will reduce the rate of childhood overweight (BMI≥85%) at age 24 months.

ELIGIBILITY:
Specific Inclusion Criteria at the parent-child dyad level will include:

* Consent from a primary caregiver (i.e., parent or legal guardian)
* Caregiver's ability to speak English or Spanish
* Infant presenting for a 2 month well-child visit (child is 6 ≥ 12 weeks old)
* Caregiver agrees to participate in the study, and agrees to bring their child to all well-child care visits until their 2 year well-child care visit.

Specific Exclusion Criteria at the parent-child dyad level will include:

* Child born prior to 32 weeks' gestational age or with a birth weight < 1500 grams
* Child with weight/length < 3rd percentile at 2 months of age
* Child with a diagnosis of failure to thrive or with weight that has dropped ≥ 2 percentile curves since the previous well child visit
* Child with known medical problems that may affect their ability to thrive or requires a special diet (e.g. metabolic disease, uncorrected congenital heart disease, renal disease, lung disease)
* Caregiver with significant mental or neurologic illness likely to impair their ability to participate
* Caregiver age < 18 years
* Caregiver with known plans to move out of the immediate area during the study period
* Caregiver with poor visual acuity (i.e. vision worse than 20/50 with Rosenbaum Pocket Screener as assessed at the time of recruitment)

Specific Inclusion Criteria at the Pediatric Resident level will include:

* Participation in the medical center's pediatric resident training program
* Providing regular care (> 3 sessions per month) in the pediatric resident primary care clinic; AND
* Consent to participate in the study

Specific Exclusion Criteria at the Pediatric Resident level will include:

* Providing no regular care in the pediatric resident primary care clinic (e.g., transitional-year resident, Medicine/Pediatrics resident); OR
* Known plans to leave the training program during the ensuing 6 months

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 865 (Actual)
Dates: Start 2010-04-28 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
Percent of children overweight or obese (BMI ≥ 85th%) at 2 years of life | 2 years

SECONDARY OUTCOMES:
BMI z score | 2 years
Change in Weight/Length z-score over time | 2 years
Parental report of infant eating and physical activity behaviors | assessed at each well child visit
Parental assessment of physician communication | each clinic visit
Parental self-efficacy | 2 years
Physician knowledge and satisfaction | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Russell L Rothman, MD MPP, Principal Investigator — Vanderbilt University; Lee Sanders, MD MPH, Principal Investigator — Stanford University; Kori Flower, MD MS MPH, Principal Investigator — UNC Chapel Hill; Shonna Yin, MD MS, Principal Investigator — NYU; Alan Delamater, LP PhD, Principal Investigator — University of Miami; Eliana Perrin, MD MPH, Principal Investigator — Duke University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Sanders LM, Perrin EM, Yin HS, Delamater AM, Flower KB, Bian A, Schildcrout JS, Rothman RL; Greenlight Study Team. A Health-Literacy Intervention for Early Childhood Obesity Prevention: A Cluster-Randomized Controlled Trial. Pediatrics. 2021 May;147(5):e2020049866. doi: 10.1542/peds.2020-049866. PMID 33911032
- [Derived] Schilling S, Ritter VS, Skinner A, Yin HS, Sanders LM, Rothman RL, Delamater AM, Perrin EM. Relationship Between Parental Locus of Control and Childhood Injury. J Prim Prev. 2020 Dec;41(6):547-565. doi: 10.1007/s10935-020-00615-y. Epub 2020 Oct 26. PMID 33104944
- [Derived] Heerman WJ, Perrin EM, Sanders LM, Yin HS, Coyne-Beasley T, Bronaugh AB, Barkin SL, Rothman RL. Racial and Ethnic Differences in Injury Prevention Behaviors Among Caregivers of Infants. Am J Prev Med. 2016 Oct;51(4):411-8. doi: 10.1016/j.amepre.2016.04.020. Epub 2016 Jun 9. PMID 27291075
- [Derived] Wood CT, Skinner AC, Yin HS, Rothman RL, Sanders LM, Delamater AM, Perrin EM. Bottle Size and Weight Gain in Formula-Fed Infants. Pediatrics. 2016 Jul;138(1):e20154538. doi: 10.1542/peds.2015-4538. Epub 2016 Jun 7. PMID 27273748
- [Derived] Brown CL, Skinner AC, Yin HS, Rothman RL, Sanders LM, Delamater AM, Ravanbakht SN, Perrin EM. Parental Perceptions of Weight During the First Year of Life. Acad Pediatr. 2016 Aug;16(6):558-64. doi: 10.1016/j.acap.2016.03.005. Epub 2016 Mar 19. PMID 27002214
- [Derived] Sanders LM, Perrin EM, Yin HS, Bronaugh A, Rothman RL; Greenlight Study Team. "Greenlight study": a controlled trial of low-literacy, early childhood obesity prevention. Pediatrics. 2014 Jun;133(6):e1724-37. doi: 10.1542/peds.2013-3867. Epub 2014 May 12. PMID 24819570
- [Derived] Perrin EM, Rothman RL, Sanders LM, Skinner AC, Eden SK, Shintani A, Throop EM, Yin HS. Racial and ethnic differences associated with feeding- and activity-related behaviors in infants. Pediatrics. 2014 Apr;133(4):e857-67. doi: 10.1542/peds.2013-1326. Epub 2014 Mar 17. PMID 24639273